CLINICAL TRIAL: NCT06747013
Title: Treatment of Focal Ventricular Tachycardias Using a Pulsed Field Ablation From a Point Ablation Catheter Short Title FOCUS-PFA
Acronym: FOCUS PFA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vivek Reddy (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor-Investigator, Vivek Reddy, Director Arrhythmia Service MSHS, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-24-00971
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Focal Ventricular Arrhythmias; Premature Ventricular Contractions; Ventricular Tachycardias
Keywords: Ventricular Arrhythmias; PVCs; Premature Ventricular Contractions; VT; Ventricular Tachycardias; Symptomatic Sustained Monomorphic Ventricular Tachycardia
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: single-arm clinical pilot study; all patients will undergo a standard ablation protocol using the study catheter (Farapoint).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ablation using study catheter (Experimental): All patients will undergo a standard ablation protocol using the study catheter (Farapoint)
  Interventions: Device: Point Ablation Catheter

INTERVENTIONS:
Device: Point Ablation Catheter — a point ablation catheter using a pulse field energy
  Other Names: Farapoint

SUMMARY:
The purpose of this study is to examine the use of a point ablation catheter (Farapoint, Boston Scientific) in the mapping and ablation of focal ventricular arrhythmias (premature ventricular contractions or ventricular tachycardia) using pulsed field energy.

DETAILED DESCRIPTION:
Study Design - This is a prospective, single-center, single-arm clinical pilot study to assess the safety and effectiveness of ablation of focal ventricular arrhythmias using the Farapoint catheter.

Sample Size - A total of 30 subjects will be included in this study. All patients will undergo treatment with the study PFA catheter.

Study Population - The target population is subjects who are planned to undergo a clinically-indicated ablation procedure for managing their focal ventricular arrhythmias - premature ventricular contractions or ventricular tachycardias.

Study Duration - Approximately 12 months: 3 months site start-up, 6 months enrollment and 3 months of follow up.

Participant Duration - Subjects will undergo brief pre-procedural testing, the ablation procedure, and 3 months of post-procedural follow up.

Primary Effectiveness Endpoint Chronic Single-Procedure Success: defined as a reduction in the burden of premature ventricular contracts (>80%) for patients treated for PVCs or absence of sustained focal ventricular tachycardia for patients being treated for focal VTs without an increase in anti-arrhythmic medications at 3 month follow ups.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet ALL of the following inclusion criteria to be eligible for participation in this clinical investigation:

* Patient is planned for a catheter ablation procedure to ablate either:

  * Premature ventricular contractions (PVCs) and a class I or IIa indication for catheter ablation of PVCS according to the 2019 HRS/EHRA/APHRS/LAHRS guidelines
  * Symptomatic Sustained Monomorphic Ventricular Tachycardia
* Able and willing to provide written consent and comply with all testing and follow-up requirements
* Above 18 years of age

Exclusion Criteria:

* Documented intracardiac thrombus or (if this can be dissolved with anticoagulation, the patient would then be eligible to participate)
* Contraindication to anticoagulation
* Life expectancy or other disease processes likely to limit survival to less than 12 months.
* Currently enrolled in an investigational study evaluating another device, biologic, or drug, that would interfere with this trial.
* NYHA Class IV heart failure
* Severe, untreated coronary artery disease which would preclude infusion of provocative agents
* Severe aortic stenosis (AVA < 1.0cm, or PG > 64mmHg)
* Severe mitral regurgitation.
* Allergy to contrast which is unable to be adequately pre-medicated.
* Acute non-cardiovascular illness or systemic infection
* Thrombocytopenia (platelet count < 50,000/mm3) or coagulopathy unless corrected
* Cardiogenic shock unrelated to ventricular arrhythmias
* Pregnancy or anticipated pregnancy during study follow-up
* PVCs or VT, which are felt to be secondary to electrolyte imbalances active thyroid disease or any reversible non-cardiac cause.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Freedom from PVC/VT recurrence | at 3 months following ablation procedure
  Freedom from PVC/VT recurrence defined as a reduction in the burden of premature ventricular contracts (>80%) for patients treated for PVCs or absence of sustained focal ventricular tachycardia for patients being treated for focal VTs without an increase in anti-arrhythmic medications at 3 month follow ups.
  (Sustained Focal Tachycardia is defined as that persisting for > 30 seconds or ventricular tachycardia which is sufficient to result in hemodynamic effect (i.e. hypotension or syncope))

SECONDARY OUTCOMES:
Incidence of Adverse events | at 3 months following ablation procedure
  Safety is measured as incidence of Serious Adverse Device Effects (SADEs)
Incidence of Serious Adverse Events (SAEs) | at 3 months following ablation procedure
  Safety is measured as incidence of Serious Adverse Events (SAEs)
Incidence of non-serious adverse events | at 3 months following ablation procedure
  Safety is measured as incidence of non-serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No